CLINICAL TRIAL: NCT04764253
Title: Examining the Individual Response to a Restricted Sodium Diet in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20200504H; KL2TR002646 (NIH)
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Sodium Watcher Program + Digital Self-Monitoring (Experimental)
  Interventions: Behavioral: Modified Sodium Watcher Program + Digital Self-Monitoring
- Usual care + Digital Self-Monitoring (Active Comparator)
  Interventions: Behavioral: Usual care + Digital Self-Monitoring

INTERVENTIONS:
Behavioral: Modified Sodium Watcher Program + Digital Self-Monitoring — Participants randomized to the experimental group will be asked to follow the modified Sodium Watchers Program intervention along with goal setting for low salt foods. Each participant will be registered to assign a unique ID in the Connected Health Platform developed by the Center on Smart and Connected Health Technologies at UT Health Science Center San Antonio and each account from the individuals' wireless and wearable devices (Fitbit and BP monitor) will be connected to his or her unique ID through this platform. Participants will be instructed to log their activities in real-time, including food intake and in-home BP monitoring using Fitbit and accompanied mobile app and BP monitor. Through the Connected Health Platform, the Fitbit app and BP monitor will transmit the data of the intervention group to the research team.
  Arms: Modified Sodium Watcher Program + Digital Self-Monitoring
Behavioral: Usual care + Digital Self-Monitoring — Participants randomized to the control group will be asked to follow usual care which is based on their routine medical and nursing care for hypertension that consists of a recommendation to follow a sodium-restricted diet and take medications as prescribed. The participants will receive wireless and wearable devices (Fitbit wristband, BP monitor). Each participant will be registered to assign a unique ID in the Connected Health Platform at the baseline and each account from the individual's wireless and wearable devices (Fitbit and BP monitor) will be connected to their unique ID through this platform. Participants will be instructed to log their activities in real-time, including food intake and in-home BP monitoring using Fitbit and accompanied mobile app and BP monitor.
  Arms: Usual care + Digital Self-Monitoring

SUMMARY:
Excessive dietary sodium intake is an independent risk factor for hypertension and cardiovascular disease. A vast array of efforts have tried to reduce sodium consumption based on evidence indicating a public health benefit. Yet this benefit has been questioned, mainly based on studies showing variability in individual responses to a sodium-restricted diet (SRD). The effects of an SRD on blood pressure vary, and adherence to an SRD is not optimal. The original Sodium Watchers Program (R01NR012967) was developed and implemented by Dr. Misook Chung (University of Kentucky). In this pilot study, the modified Sodium Watchers Program will propose improving adherence to an SRD through education and digital self-monitoring for daily sodium intake and blood pressure.

In addition, few studies have examined individuals' metabolic responses to the SRD. In a secondary analysis, we further will examine genetic variants associated with salt sensitivity and whether such a genetic component is associated with sodium excretion and BP control.

A total of 40 hypertensive patients will be randomly assigned to the intervention (n=20) or control group (n=20). The intervention group will receive 8-week education sessions remotely using a video conferencing program. All participants will collect a 24-hour urine specimen for sodium excretion and a total of 4.0ml of peripheral blood will be drawn for salt sensitivity during baseline visit. All participants will be asked to log their activities in real-time, including food intake and in-home BP monitoring using Fitbit and accompanied mobile app and BP monitor.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure of 120-159 mmHg or diastolic blood pressure of 80-99 mmHg, whether or not taking blood pressure medications.
* Smartphone with a data plan
* Valid email address
* Willing and able to participate in online study videoconferencing visits (Zoom)
* Reads and writes in English

Exclusion Criteria:

* Participating in another related research study
* Cardiovascular disease event (e.g. stroke, myocardial infarction) in prior 6 months
* Active cancer
* Recent hospitalization due to psychiatric condition or event
* Pregnancy or breastfeeding - current or planned during the study period
* Documented dementia
* Prisoners
* Diabetes Diagnosis
* Heart Failure Diagnosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure over time | Up to 8 weeks
  Blood pressure (BP) will be measured using a Vital Signs Monitor 300 Series model (WelchAllyn, US). The midsection circumference of the dominant upper arm will be measured with a tape measure, and the proper sized cuff will be selected accordingly. Systolic and diastolic BP will be measured in the dominant arm twice with a 2-minute rest period between measures; two measures will be averaged.
Change in adherence to sodium restricted diet over time | Up to 8 weeks
  Participants will complete a 24-hour urinary sodium excretion test at baseline and at 8 weeks after the intervention is completed. 24-hour urinary sodium excretion (mg excreted/day) will be tested by collecting all urine excreted over 24 hours. Participants are asked to note the time when they start in a written log, then discard the first urine after that time. They will then collect all urine excreted over the course of the next 24 hours, noting down the time and amount excreted each time in the written log. Urine is stored in a container and does not need refrigeration. 24-hour urine sodium samples will be analyzed by the Center for Renal Precision Medicine laboratory.

SECONDARY OUTCOMES:
Adherence to dietary sodium intake monitoring | Up to 8 weeks
  Adherence to dietary sodium intake monitoring will be monitored using Fitbit companion mobile dietary app. The Fitbit app is intended as an intervention tool to enhance self-monitoring and promote adherence, not a reliable assessment tool for dietary sodium intake (24-hour urinary samples will be used for that purpose as described in outcomes section). Each subject will be registered to assign a unique ID in the platform developed by the Center on Smart and Connected Health Technologies at UT Health San Antonio, and each account from the individuals' Fitbit will be connected to his or her unique ID through this platform. Subjects will be instructed to log their food intake in real-time. Percentage of days that subject log his or her meal in the dietary app with a calorie intake of over 1000 will be used to measure adherence to dietary sodium intake monitoring.
Adherence to In-home BP monitoring | Up to 8 weeks
  Adherence to In-home BP monitoring will be measured by the percentage of days that subject log in-home BP using a wireless and automatic BP monitor device (Omron 7 Series Upper Arm BP Monitor). It has a range of 0 to 299 mmHg for BP and 40 to 180 beats per minute (bpm) for heart rate (HR). The cuff is inflated using an electric pump and deflated by means of a pressure release valve. After each measurement, the SBP, DBP, and HR are shown on the LCD screen. The device can also display a symbol on the screen indicating an irregular heartbeat detected during measurement of SBP and DBP. Each subject will be registered to assign a unique ID in the Connected Health Platform and each account from the individuals' Omron mobile app will be connected to his or her unique ID through this platform. Subjects will be instructed to measure BP while in a sitting position and transfer the BP data to Omron mobile app using a wireless and automatic BP monitor device.
Attendance at education sessions | Up to 8 weeks
  Attendance at education sessions will be measured by number of attended sessions for the 8-week education sessions in intervention group.
Retention rate | Up to 8 weeks
  Retention rate will be measured by the percentage of subjects who come to the follow-up visit (8 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Jisook Ko, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this time.

REFERENCES:
- [Derived] Ko J, Wang J, Chung ML, Sharma K. Examining the Individual Response to a Low-Sodium Diet in Patients with Hypertension: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Feb 13;12:e39058. doi: 10.2196/39058. PMID 36780210

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT04764253/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT04764253/ICF_001.pdf